CLINICAL TRIAL: NCT07207551
Title: Prevalence of Hb Variants and Haemoglobinopathies in a Tertiary Care Hospital: A Retrospective Cross-sectional Study
Brief Title: Prevalence of Hemoglobinopathies Associated With Significant Hb Variants in the Chattogram Region of Bangladesh
Acronym: Hb variants
Status: Completed | Type: Observational
Sponsor: Bangladesh Bioscience Research Group (Network)
Responsible Party: Principal Investigator, Pair Ahmed Jiko, Lab-Incharge (Biochemist), Chittagong Medical College
Other Study IDs: BBMH/2024/RP-2412; BBMH/January/2024/024 (Other: Institute of Applied Health Sciences Hospital-USTC (Ex: BBMH))
Record Dates: First submitted 2025-09-14; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Hemoglobinopathies
Keywords: Hb Variants; HbE Trait; Beta Thalassemia; Iron Profile; Peripheral Blood Film (PBF)
MeSH Terms: conditions — Hemoglobinopathies; beta-Thalassemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hemoglobinopathies represent a collection of genetic conditions that influence the structure or synthesis of haemoglobin, the protein found in red blood cells that facilitates oxygen transport from the lungs throughout the body. This research proposal presents a study evaluating the prevalence of hemoglobinopathies and their significant haemoglobin variants within a specific population. The research will employ a cross-sectional study design, recruiting participants through community outreach efforts and healthcare facilities while obtaining informed consent. Data will be collected with the utmost precision and rigor, using advanced screening techniques such as high-performance liquid chromatography (HPLC), capillary electrophoresis, and molecular analysis. The gathered data will be processed to assess haematological parameters, including RBC, Iron Ferritin, TIBC, electrophoresis profiles (HbA, HbA2, HbE, HbF), MCV, MCHC, and PCV among individuals with hemoglobinopathies (HbE disease/trait, Beta thalassemia disease/trait, heterozygous HPFH, HbE-beta thal). They will examine variations relative to demographic factors. The expected results will have substantial clinical and public health consequences by enhancing genetic counselling, informing clinical decision-making, and strengthening public health initiatives.

DETAILED DESCRIPTION:
Hemoglobinopathies are genetic disorders affecting the structure or production of hemoglobin, the oxygen-carrying protein in red blood cells. This study aims to determine the prevalence and major variants of hemoglobinopathies in a target population using a cross-sectional design. Participants will be recruited through community outreach and healthcare facilities with informed consent. Screening will involve advanced techniques such as HPLC, capillary electrophoresis, and molecular analysis, alongside hematological assessments (RBC, ferritin, TIBC, MCV, MCHC, PCV, and hemoglobin profiles: HbA, HbA2, HbE, HbF). Findings will be analyzed in relation to demographic factors.

ELIGIBILITY:
Inclusion Criteria:

* Residents of the Chattogram metropolitan area.
* All ages and both sexes with informed consent.
* Willing to provide venous blood samples.
* No blood transfusion in the past 3 months.

Exclusion Criteria:

* Refusal or withdrawal of consent.
* Blood transfusion within the last 3 months.
* Pregnant women.
* Inadequate or hemolyzed blood samples.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population will consist of individuals from the selected community and healthcare facilities who meet the inclusion criteria. Participants of all ages and both sexes will be included, provided they give informed consent and have not received a blood transfusion within the last three months. The population is expected to represent a cross-section of healthy individuals and those with suspected or confirmed hemoglobinopathies, allowing for assessment of hemoglobin variants and related biochemical parameters.
Sampling Method: Non-Probability Sample
Enrollment: 760 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-09-04 (Actual)

PRIMARY OUTCOMES:
Detection of Hemoglobin Variants by Hb-Electrophoresis | Day 1, at enrollment
  Performed to detect hemoglobin variants (e.g., HbA, HbE, HbS, HbC, HbD, HbF). The outcome will report the number and percentage of participants with each variant.

SECONDARY OUTCOMES:
Correlation of Hematological Parameters with Demographic Factors | Day 1, upon enrollment
  Statistical correlation between hematological indices and demographic factors (eg. age, sex, family history).

CONTACTS AND LOCATIONS:
Overall Officials: PAIR AHMED JIKO, Lab-Incharge (Biochemist), Principal Investigator — Institute Of Applied Health Sciences Hospital-USTC (Ex-BBMH)
Locations (1):
- University of Science and Technology Chittagong (USTC), Khulshi, Chattogram, Bangladesh

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared with other researchers to protect patient confidentiality and comply with institutional and ethical guidelines. Only aggregated, de-identified data may be shared upon reasonable request and with appropriate ethical approvals.